CLINICAL TRIAL: NCT05969275
Title: Umbilical Mesenchymal Stromal Cells as Cellular Immunotherapy for Septic Shock: A Multi-Center, Double Blind, Phase II Randomized Controlled Trial
Brief Title: Umbilical Mesenchymal Stromal Cells as Cellular Immunotherapy for Septic Shock
Acronym: UC-CISSII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Stem Cell Network (Other); Canadian Critical Care Trials Group (Other); Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UC-CISSII
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Septic Shock; Sepsis; Pathologic Processes; Shock; Systemic Inflammatory Response Syndrome; Inflammation; Infections
Keywords: Mesenchymal Stem Cells; Mesenchymal Stromal Cells; Randomized Controlled Trial; Cryopreserved; Allogeneic; Umbilical Cord; Phase II; Sepsis; Septic Shock
MeSH Terms: conditions — Shock, Septic; Sepsis; Pathologic Processes; Shock; Systemic Inflammatory Response Syndrome; Inflammation; Infections

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Mesenchymal Stromal Cells (UC-MSCs) (Experimental): Intravenous infusion of 300 million allogeneic, cryopreserved, umbilical cord-derived human mesenchymal stromal cells
  Interventions: Biological: Allogeneic umbilical cord-derived human mesenchymal stromal cells
- Placebo (Placebo Comparator): Intravenous infusion of placebo, with excipients
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogeneic umbilical cord-derived human mesenchymal stromal cells — Intravenous infusion of 300 million allogeneic, cryopreserved, umbilical cord-derived human mesenchymal stromal cells
  Arms: Umbilical Cord Mesenchymal Stromal Cells (UC-MSCs)
Other: Placebo — Intravenous infusion of placebo, with excipients
  Arms: Placebo

SUMMARY:
Septic shock is associated with substantial burden in terms of both mortality and morbidity for survivors of this illness. Pre-clinical sepsis studies suggest that mesenchymal stem (stromal) cells (MSCs) modulate inflammation, enhance pathogen clearance and tissue repair and reduce death. Our team has completed a Phase I dose escalation and safety clinical trial that evaluated MSCs in patients with septic shock. The Cellular Immunotherapy for Septic Shock Phase I (CISS) trial established that MSCs appear safe and that a randomized controlled trial (RCT) is feasible. Based on these data, the investigators have planned a phase II RCT (UC-CISS II) at several Canadian academic centres which will evaluate intermediate measures of clinical efficacy (primary outcome), as well as biomarkers, safety, clinical outcome measures, and a health economic analysis (secondary outcomes).

DETAILED DESCRIPTION:
Septic shock is a devastating illness and the most severe form of infection seen in the intensive care unit (ICU). It is characterized by cardiovascular collapse, failure of organs and is common with severe repercussions including a mortality of 20-40%. Survivors suffer long-term impairment in function and reduced quality of life (QOL). Despite decades of research examining different immune therapies, none has proven successful and supportive care remains the mainstay of therapy, at a cost of approximately 4-billion dollars in Canada annually. MSCs represent a potentially novel treatment for sepsis because in animal models, MSCs have been shown to modulate the immune system, increase pathogen clearance, restore organ function, and reduce death.

The Phase II multi-centre double blind Umbilical Cord Cellular Immunotherapy for Septic Shock RCT (UC-CISS II) will examine intermediate measures of clinical efficacy (primary outcome) as well as biomarkers, safety, clinical outcome measures, and a health economic analysis (secondary outcomes). To answer these aims, UC-CISS II will randomize 296 patients who are admitted to the ICU with septic shock to 300 million cryopreserved, allogeneic, umbilical cord-derived MSCs or placebo across several Canadian academic centres over approximately 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all the following inclusion criteria at time of randomization to be eligible:

1. At least 18 years of age AND
2. Requirement for admission to the intensive care unit AND
3. Index admission to the intensive care unit AND
4. Cardiovascular organ failure for at least 1 consecutive hour defined by the requirement of at least 5 mcg/min of norepinephrine or 100 mcg/min of phenylephrine or 0.03 U/min vasopressin AND
5. Clinician impression that cardiovascular organ failure is related to infection AND
6. There is at least 1 other acute organ failure according to modified individual Sequential Organ Failure Assessment Scores within 24 hours of meeting Cardiovascular organ failure defined by:

   1. Respiratory failure: invasive or non-invasive mechanical ventilation with a positive end expiratory pressure (PEEP) >/= 5 cm H2O and a partial pressure of oxygen/fractional inspired oxygen concentration (P/F ratio </= 200), OR high-flow nasal canula oxygen therapy (minimum total flow rate of 30 lpm and 40% FiO2); OR
   2. Hematological failure: platelet count of </= 100 X 10^9/L OR
   3. Acute kidney injury: acute renal insufficiency with a creatinine of >/= 200 umol/L, or the requirement for new renal replacement therapy, or for participants with known chronic renal failure but not on dialysis, a 50% increase in their baseline creatinine concentration OR
   4. Organ hypoperfusion: a lactate >/= 4 mmol/L

Acute organ failures that meet eligibility criteria must not have been present for greater than 48 hours prior to meeting the eligibility criteria.

Exclusion Criteria:

Patients will be excluded if they have at least one of the following at time of randomization:

1. Another form of shock (cardiogenic, hypovolemic, obstructive) OR
2. History of known chronic pulmonary hypertension with a WHO functional class of IV OR
3. History of severe chronic pulmonary disease requiring home oxygen OR
4. History of severe chronic cardiac disease including congestive heart failure or valvular dysfunction with a New York Heart Association Functional class IV or severe chronic ischemic heart disease with a Canadian Cardiovascular Society angina class score IV OR
5. History of severe chronic liver disease (Child-Pugh Class C or model for end stage liver disease (MELD) Score >= 15) OR
6. Malignancy in previous 1 year (excluding resolved non-melanoma skin cancer) OR
7. Treating physician impression that death is imminent within the 12 hours after meeting eligibility criteria OR
8. Pregnant or lactating OR
9. Family or patient not committed to aggressive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Days free from mechanical ventilation and/or vasopressors and/or renal replacement therapy | Through to 28 days post-randomization
  The number of days free from each of these support measures

SECONDARY OUTCOMES:
Biomarkers - Vascular permeability | At baseline, 1, 3 and 7 days post-randomization
  Markers of vascular permeability (ex: Angpt1 and 2)
Biomarkers - Acute kidney injury | At baseline, 1, 3 and 7 days post-randomization
  Markers of acute kidney injury (ex: Urine TIMP2-IGFBP7, IL-18)
Biomarkers - Muscle weakness | At baseline, 1, 3 and 7 days post-randomization
  Markers of muscle weakness (ex: micro RNA [miR] miR-181a, growth differentiation Factor-15)
Biomarkers - Pathogen clearance | At baseline, 1, 3 and 7 days post-randomization
  Mechanisms related to pathogen clearance (ex: cathelicidin, LL-37)
Biomarkers - Inflammatory mediators and cytokines | At baseline, 1, 3 and 7 days post-randomization
  Pro- and anti-inflammatory mediators and cytokines (ex: CRP, IL-6, IL-8, IL-10, IL-1B and IL1-RA)
Safety - Adverse Event | Through to 7 days post-randomization
  Safety of study treatment administration, examined for the occurrence of any adverse event (which requires treatment or intervention) regardless of relationship to study treatment
Safety - Serious and Unexpected Adverse Events | Through to 28 days post-randomization
  Safety of study treatment administration, examined for the occurrence of serious and unexpected adverse events that are considered possibly or related to the study treatment
Safety - Expected Adverse Events | Through to 28 days post-randomization
  Safety of study treatment administration, examined for the occurrence of expected adverse events (including nosocomial infections, acute coronary syndrome, tachy and bradyarrhythmia, clinically important bleeding, ARDS and thrombotic/thromboembolic events)
Mortality | In ICU (through study completion, up to 1 year), in hospital (through study completion, up to 1 year), 28 days, 90 days, 6 months and 1 year post-randomization
  All-cause mortality
Length of ICU Stay (in days) | Number of elapsed days from admission until ICU discharge, up to 1 year
  Time in ICU
Length of Hospital Stay (in days) | Number of elapsed days from admission until hospital discharge, up to 1 year
  Time in hospital
Hospital Re-Admissions | At 28 days, 90 days and 1 year post-randomization
  Re-admission to any hospital
ICU Re-Admissions | During index study hospital admission (through study completion, up to 1 year)
  Re-admission to ICU during study hospital admission
Organ Failure Rates | Through to 90 days post-randomization
  Organ failure rates (using Sequential Organ Failure Assessment Score), described individually and in composite
Days free from mechanical ventilation | Through to 90 days post-randomization
  Number of days free from mechanical ventilation
Days free from vasopressors | Through to 90 days post-randomization
  Number of days free from vasopressor agents
Days free from renal replacement therapy | Through to 90 days post-randomization
  Number of days free from renal replacement therapy
Patient Reported Outcomes - Functional Independence Measure (FIM) | At 30 days, 6 months and 1 year post-randomization
  FIM scores ranging from 18 to 126 (where the higher the score, the more independent the patient is)
Patient Reported Outcomes - Short Form Survey-36 (SF-36) | At 30 days, 6 months and 1 year post-randomization
  SF-36 scores ranging from 0 to 100 (with higher scores indicating better health status)
Health Economic Analysis | Through to 28 days post-randomization
  A cost-utility analysis of MSCs compared to placebo from a perspective of Canada's publicly funded health care system will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Lauralyn McIntyre, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital (General Campus), Ottawa, Ontario
  - The Ottawa Hospital (Civic Campus), Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No